CLINICAL TRIAL: NCT01701856
Title: Natalizumab De-escalation to Interferon-beta-1b in Patients With Relapsing-remitting Multiple Sclerosis: A Swiss Multicenter Study Prospective, Controlled, Single-arm, Open-label, Multi-centre, Phase IV Study
Brief Title: Natalizumab De-escalation to Interferon-beta-1b in Patients With Relapsing-remitting Multiple Sclerosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Problems to recruit the needed number of patients in the planned time
Sponsor: Claudio Gobbi (Other Government)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Claudio Gobbi, Dr. med., Ospedale Civico, Lugano
Organization: Ospedale Civico, Lugano (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EOC.NSI.11.01
Record Dates: First submitted 2012-09-18; First posted 2012-10-05 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: relapsing-remitting multiple sclerosis; natalizumab; de-escalation; interferon beta-1b
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interferon beta-1b (Experimental): Interferon beta-1b 250 mcg s.c. every other day
  Interventions: Drug: Interferon beta-1b

INTERVENTIONS:
Drug: Interferon beta-1b — 250 mcg, s.c., each other day for 12 months
  Other Names: Betaferon®

SUMMARY:
Multiple Sclerosis (MS) is the most common neurological disorder causing disability in young adults affecting approximately 1 in 1.000 people in western countries. The clinical manifestations usually begin at the age of 20 to 40 years with a median age of 28 years at onset with acute episodes of neurological dysfunction, followed by periods of partial or complete remission and clinical stability in between relapses. This relapsing-remitting phase (RR-MS) of the disease is usually followed by progressive clinical disability (secondary progressive phase, SP-MS).

At present, there is no cure for MS. Based on the pathological concept that neuroinflammation is the common element leading or contributing to neurodegenerative changes, immune interventions have been introduced into clinical practice such as Natalizumab (Tysabri), a humanized monoclonal antibody. Natalizumab (Tysabri) is indicated as a disease-modifying monotherapy of highly active relapsing MS. The associated risks, especially progressive multifocal leukoencephalopathy, necessitate active monitoring of patients and a continuous discussion of optimum use of this drug. In clinical practice, the question how to manage patients on natalizumab at a higher risk for progressive multifocal leukoencephalopathy remains unresolved.

This prospective, controlled (comparison to the period prior to natalizumab treatment), single-arm, open-label, multi-centre, phase IV study aims to evaluating the concept of natalizumab de-escalation to interferon-beta-1b e.o.d in relapsing-remitting multiple sclerosis patients, who consider stopping natalizumab due to a benefit-risk assessment. In particular, to evaluating if interferon beta-1b treatment may be able to overcome the recurrence of significant clinical and radiological disease activity after natalizumab cessation and may keep disease activity better under control as compared to the time prior to natalizumab.

The study population includes patients with relapsing-remitting multiple sclerosis (RR-MS) being treated at least for 12 months with natalizumab and having decided to stop natalizumab treatment and to de-escalate their therapy to a first line treatment with interferon beta-1b. They will be treated during 12 months with interferon-beta 1b 250 mcg given subcutaneously every other day. A 12-month follow-up period with the same treatment is planned.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients with relapsing-remitting forms of multiple sclerosis (according to McDonald's criteria);
* Age between 18 and 70 years;
* Natalizumab-treatment for at least 12 months following the current Swiss guidelines for treatment initiation;
* Treated with a disease-modifying therapy other than interferon beta-1b for at least 12 months before natalizumab was initiated;
* Never treated with interferon beta-1b;
* Eligible patients are clinically stable (free from relapses and 6-month confirmed disability progression for at least 6 months) while on natalizumab-treatment and do not show any Gd-enhancement on their last MRI performed while on Tysabri;
* In eligible patients MRI were performed in the past as following

  * 6-18 months prior to natalizumab-treatment
  * at natalizumab start
  * 12 months after natalizumab initiation;
* Good records with regard to clinical disease activity (relapse rate, EDSS progression) in the year prior to natalizumab and during natalizumab;
* Patients who decide to stop natalizumab treatment after a careful benefit/risk assessment. Risk for PML increases with duration of natalizumab exposure, pre-treatment with an immunosuppressant agent or serological status of anti-JC-virus positivity;
* Patients, who in context with cessation of natalizumab have decided, after a careful benefit/risk assessment, to continue treatment of their MS with Interferon beta-1b;
* Women of potential childbearing with active contraceptive methods;
* Patients who are willing to undergo study procedures;
* Patients who are willing to undergo MRI;
* Patients who are willing and able to sign informed consent.

Exclusion Criteria:

* Patients who have previously entered this study;
* Natalizumab-treatment for less than 12 months following the current Swiss guidelines for treatment initiation;
* Prior treatment with interferon beta-1b (ever interferon beta-1b);
* Sign of clinical disease activity within the 6 months;
* One or more relapses and/or 6-month confirmed disability progression during the 6 months prior to the study;
* Secondary progressive MS;
* Primary progressive MS;
* Pregnancy - Serum pregnancy test at screening visit positive- or breast feeding;
* Uncontrolled, clinically significant heart diseases, such as arrhythmias, angina, or uncompensated congestive heart failure;
* History of severe depression or attempted suicide or current suicidal ideation;
* Medical or psychiatric conditions that compromise the ability to give informed consent, to comply with the protocol, or to complete the study;
* Uncontrolled seizure disorder;
* Myopathy or clinically significant liver disease;
* Inability, in the opinion of the principal investigator or staff, to comply with protocol requirements for the duration of the study;
* Known hypersensitivity to interferon-beta or other human proteins including albumin;
* Any contraindication for MRI or contrast administration;
* A history of drug abuse in the 6 months prior to screening;
* Treatment with any of the following in the 30 days before day 1: systemic corticosteroids, ACTH, or other investigational drugs;
* Participation in any other study involving investigational or marketed products, concomitantly or within 30 days prior to entry in the study;
* Current participation on other clinical trials;
* Treatment with drugs which might interfere with the evaluation of study drugs during the study protocol such as immunomodulants, immunosuppressives other than interferon beta-1b;
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol such as immunomodulants, immunosuppressives other than interferon beta-1b.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Annualized relapse rate on study compared to annualized relapse rate in the year prior to natalizumab initiation on first line disease modifying treatment (month -24 to -12) | 12 months
Annualized relapse rate on study compared to annualized relapse rate in the year prior to natalizumab initiation on first line disease modifying treatment (month -24 to -12) | 3 months
Annualized relapse rate on study compared to annualized relapse rate in the year prior to natalizumab initiation on first line disease modifying treatment (month -24 to -12) | 6 months
Annualized relapse rate on study compared to annualized relapse rate in the year prior to natalizumab initiation on first line disease modifying treatment (month -24 to -12) | 9 months
Annualized relapse rate on study compared to annualized relapse rate in the year prior to natalizumab initiation on first line disease modifying treatment (month -24 to -12) | 15 months
Annualized relapse rate on study compared to annualized relapse rate in the year prior to natalizumab initiation on first line disease modifying treatment (month -24 to -12) | 18 months
Annualized relapse rate on study compared to annualized relapse rate in the year prior to natalizumab initiation on first line disease modifying treatment (month -24 to -12) | 21 months
Annualized relapse rate on study compared to annualized relapse rate in the year prior to natalizumab initiation on first line disease modifying treatment (month -24 to -12) | 24 months

SECONDARY OUTCOMES:
Severity of relapses | 3 months
Severity of relapses | 6 months
Severity of relapses | 9 months
Severity of relapses | 12 months
Severity of relapses | 15 months
Severity of relapses | 18 months
Severity of relapses | 21 months
Severity of relapses | 24 months
Proportion of relapse free patients | 3 months
Proportion of relapse free patients | 6 months
Proportion of relapse free patients | 9 months
Proportion of relapse free patients | 12 months
Proportion of relapse free patients | 15 months
Proportion of relapse free patients | 18 months
Proportion of relapse free patients | 21 months
Proportion of relapse free patients | 24 months
3-month confirmed EDSS progression | 3 months
  of at least 1.0 points if score < 5.5, at least 0.5 points if score ≥ 5.5
3-month confirmed EDSS progression | 6 months
  of at least 1.0 points if score < 5.5, at least 0.5 points if score ≥ 5.5
3-month confirmed EDSS progression | 9 months
  of at least 1.0 points if score < 5.5, at least 0.5 points if score ≥ 5.5
3-month confirmed EDSS progression | 12 months
  of at least 1.0 points if score < 5.5, at least 0.5 points if score ≥ 5.5
3-month confirmed EDSS progression | 15 months
  of at least 1.0 points if score < 5.5, at least 0.5 points if score ≥ 5.5
3-month confirmed EDSS progression | 18 months
  of at least 1.0 points if score < 5.5, at least 0.5 points if score ≥ 5.5
3-month confirmed EDSS progression | 21 months
  of at least 1.0 points if score < 5.5, at least 0.5 points if score ≥ 5.5
3-month confirmed EDSS progression | 24 months
  of at least 1.0 points if score < 5.5, at least 0.5 points if score ≥ 5.5
MSFC | 3 months
  Three part instrument composed of Timed-25-foot (7.62 m)-walk, 9 hole-peg-test (9 HPT), 3'' paced auditory serial addition test (PASAT).
MSFC | 6 months
  Three part instrument composed of Timed-25-foot (7.62 m)-walk, 9 hole-peg-test (9 HPT), 3'' paced auditory serial addition test (PASAT).
MSFC | 9 months
  Three part instrument composed of Timed-25-foot (7.62 m)-walk, 9 hole-peg-test (9 HPT), 3'' paced auditory serial addition test (PASAT).
MSFC | 12 months
  Three part instrument composed of Timed-25-foot (7.62 m)-walk, 9 hole-peg-test (9 HPT), 3'' paced auditory serial addition test (PASAT).
MSFC | 18 months
  Three part instrument composed of Timed-25-foot (7.62 m)-walk, 9 hole-peg-test (9 HPT), 3'' paced auditory serial addition test (PASAT).
MSFC | 21 months
  Three part instrument composed of Timed-25-foot (7.62 m)-walk, 9 hole-peg-test (9 HPT), 3'' paced auditory serial addition test (PASAT).
MSFC | 24
  Three part instrument composed of Timed-25-foot (7.62 m)-walk, 9 hole-peg-test (9 HPT), 3'' paced auditory serial addition test (PASAT).
Change of EDSS score compared to change in the year prior to natalizumab treatment (month -24 to-12 | 3 months
Change of EDSS score compared to change in the year prior to natalizumab treatment (month -24 to-12 | 6 months
Change of EDSS score compared to change in the year prior to natalizumab treatment (month -24 to-12 | 9 months
Change of EDSS score compared to change in the year prior to natalizumab treatment (month -24 to-12 | 12 months
Change of MSFC score compared to change in the year prior to natalizumab treatment (month -24 to-12 | 3 months
Change of MSFC score compared to change in the year prior to natalizumab treatment (month -24 to-12 | 6 months
Change of MSFC score compared to change in the year prior to natalizumab treatment (month -24 to-12 | 9 months
Change of MSFC score compared to change in the year prior to natalizumab treatment (month -24 to-12 | 12 months
Number of new/enlarging T2-hyperintense lesions | 6 months
  MRI
Number of new/enlarging T2-hyperintense lesions | 12 months
  MRI
Number of new/enlarging T2-hyperintense lesions | 24 months
  MRI
Number of Gd-enhancing lesions | 6 months
  MRI
Number of Gd-enhancing lesions | 12 months
  MRI
Number of Gd-enhancing lesions | 24 months
  MRI
EQ-5D | 6 months
  Quality of life questionnaire
EQ-5D | 12 months
  Quality of life questionnaire
EQ-5D | 24 months
  Quality of life questionnaire
FAMS | 6 months
  Quality of life questionnaire
FAMS | 24 months
  Quality of life questionnaire
MSFC | 15 months
  Three part instrument composed of Timed-25-foot (7.62 m)-walk, 9 hole-peg-test (9 HPT), 3'' paced auditory serial addition test (PASAT).
EQ-5D | 18 months
  Quality of life questionnaire
FAMS | 12 months
  Quality of life questionnaire
FAMS | 18 months
  Quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Gobbi, MD, Principal Investigator — Ospedale Regionale di Lugano - Civico
Locations (1):
- Ospedale Regionale di Lugano - Civico, Lugano, Canton Ticino, Switzerland

REFERENCES:
- [Background] Multiple Sclerosis Therapy Consensus Group (MSTCG); Wiendl H, Toyka KV, Rieckmann P, Gold R, Hartung HP, Hohlfeld R. Basic and escalating immunomodulatory treatments in multiple sclerosis: current therapeutic recommendations. J Neurol. 2008 Oct;255(10):1449-63. doi: 10.1007/s00415-008-0061-1. Epub 2008 Oct 29. PMID 19005625
- [Background] Kappos L, Bates D, Edan G, Eraksoy M, Garcia-Merino A, Grigoriadis N, Hartung HP, Havrdova E, Hillert J, Hohlfeld R, Kremenchutzky M, Lyon-Caen O, Miller A, Pozzilli C, Ravnborg M, Saida T, Sindic C, Vass K, Clifford DB, Hauser S, Major EO, O'Connor PW, Weiner HL, Clanet M, Gold R, Hirsch HH, Radu EW, Sorensen PS, King J. Natalizumab treatment for multiple sclerosis: updated recommendations for patient selection and monitoring. Lancet Neurol. 2011 Aug;10(8):745-58. doi: 10.1016/S1474-4422(11)70149-1. PMID 21777829
- [Background] Kappos L, Freedman MS, Polman CH, Edan G, Hartung HP, Miller DH, Montalban X, Barkhof F, Radu EW, Metzig C, Bauer L, Lanius V, Sandbrink R, Pohl C; BENEFIT Study Group. Long-term effect of early treatment with interferon beta-1b after a first clinical event suggestive of multiple sclerosis: 5-year active treatment extension of the phase 3 BENEFIT trial. Lancet Neurol. 2009 Nov;8(11):987-97. doi: 10.1016/S1474-4422(09)70237-6. Epub 2009 Sep 10. PMID 19748319
- [Background] Putzki N, Yaldizli O, Buhler R, Schwegler G, Curtius D, Tettenborn B. Natalizumab reduces clinical and MRI activity in multiple sclerosis patients with high disease activity: results from a multicenter study in Switzerland. Eur Neurol. 2010;63(2):101-6. doi: 10.1159/000276400. Epub 2010 Jan 16. PMID 20090344
- See also: home page of the main facility — http://www.eoc.ch
- See also: home page of supporting society for MS patients in Switzerland — http://www.multiplesklerose.ch/